Study Title: Randomized controlled trial of virtual reality therapy for irritable bowel syndrome.

NCT Number: NCT06687616

**Document: Informed Consent Forms** 

Document Date: 5/13/2025

CSMC Date Effective: 1/28/2025



# CONSENT FORM FOR RESEARCH / PERMISSION FORM FOR RESEARCH\* / ASSENT FOR TEENS 13-17 YEARS OF AGE For Cedars-Sinai and Participating Affiliates<sup>1</sup>

\*This form is also a Permission Form for your child to take part in this research. In this case, "you" refers to "your child."

**Study title:** Randomized controlled trial of virtual reality therapy for irritable bowel syndrome.

**Sponsor:** National Institute of Diabetes and Digestive and Kidney Diseases

Cedars-Sinai Principal Investigator: Christopher V. Almario, MD, MSHPM

Cedars-Sinai study contact phone number: 310-423-5434

To help guide your review of this form, the main sections include:

- 1. Key Information
- 2. Purpose of the Study
- 3. Main Study Procedures
- 4. Possible Benefits from Taking Part in the Study
- 5. Possible Risks and Discomforts of the Main Research Procedures
- 6. Common Medical Procedures Performed for Research Purposes and Risks
- 7. Reasons Participation May Be Stopped by the Researchers or Sponsor
- 8. Voluntary Participation and Other Options
- 9. Confidentiality Protections
- 10. Research-Related Illness or Injury
- 11. Financial Considerations
- 12. Contact for Ouestions or Problems
- 13. Authorization for Use or Disclosure of Identifiable Health Information for Research
- 14. Signature Page

<sup>&</sup>lt;sup>1</sup> The Cedars-Sinai Affiliated Covered Entity ("ACE") is comprised of covered entities under the common ownership or control of Cedars-Sinai Health System, including Cedars-Sinai Medical Center (CSMC); Cedars-Sinai Medical Care Foundation; Cedars-Sinai Marina Del Rey Hospital (MDRH); Torrance Memorial Medical Center (TMMC); Torrance Health Association, Inc., d/b/a Torrance Memorial Physician Network; Huntington Hospital (HH), and Huntington Medical Foundation.

CSMC Date Effective: 1/28/2025

#### 1. Key Information

Thank you for considering research participation. Research helps make medical and scientific advancements possible. In this form, we are asking for your consent to take part in this research study. Taking part in this research study is voluntary.

This section provides key information about the study. Please take your time to read this entire form. Also, please ask questions before deciding whether to take part in this research study. You are welcome to talk with family, friends, and other healthcare providers before you decide.

- **Purpose:** The purpose of this study is to assess the impact of virtual reality (VR) therapy programs among patients with irritable bowel syndrome (IBS). Section 2 includes more details.
- **Duration:** Taking part in this study will last about 8 weeks.
- **Procedures:** The main things that will happen in this study are using a VR headset a couple times per week for about 10-15 minutes at a time, and taking weekly surveys delivered via email. Section 4 includes more details.
- **Benefits:** You may or may not benefit from being in this study. The possible benefits of taking part in this study include a reduction of abdominal pain and other IBS symptoms (e.g., bowel habit changes, bloating), and general improvement in mental health. Potential long-term benefits include continued improvement in abdominal pain and IBS symptoms, improved functionality, and improvements in overall physical and psychological health. This research will contribute to societal knowledge about the safety and effectiveness of VR therapy programs among patients with IBS. Section 3 includes more details.
- **Risks:** All research studies involve some risk. Risks or discomforts from this study may include minor psychological distress from questionnaires regarding health and employment status, risk of neck pain from wearing the headset, and ~5% risk of "cybersickness," presenting as short-term symptoms (e.g., headache, nausea, dizziness, feelings of anxiety) related to being in the 3-dimensional VR environments. Section 6 includes more details.
  - If you experience side effects or have problems during the study, contact the study team using the contact information on the first page of this consent form.
- **Alternatives:** You can choose not to be in the study. There may be other choices for you. These are described in Section 8 of this form.

CSMC Date Effective: 1/28/2025

• **New Information:** During the study, we may find out new information about this study. We will tell you about any important changes or new findings that may impact your decision to continue taking part in the study.

#### 2. Purpose of the Study

We are doing this study to see if using a VR therapy program can help manage or improve the symptoms of IBS.

You are being asked to take part in this research study because you are an outpatient at Cedars-Sinai Medical Center or were referred for this study by a physician at Cleveland Clinic, have been diagnosed with IBS, and experience clinically significant abdominal pain.

These VR therapy programs have not been approved by the U.S. Food and Drug Administration (FDA) because they are still being studied. The VR headset you will use is commercially available and is not being studied in this research.

The study will include up to 72 people total.

#### 3. Main Study Procedures

All participants will be provided with a Meta Quest 2 headset, which will be loaded with one of two VR programs. Both VR programs include audio and visual experiences. Participants will be asked to use the headset a couple times per week (for about 10-15 minutes at a time) for a total of 8 weeks.

You may receive text messages and email reminders as part of this study. Usual text messaging costs may apply and are not paid for by the research team. You will be responsible for these costs. You will be able to opt-out of text messages; please tell the study team if you do not want to receive text messages. You may also need to use a smartphone or computer application (app) as part of this research. The study team will help you set this up if necessary.

This is a randomized, single-blind research study. Here's a breakdown of what these words mean:

• Randomized: This means that you will be put in a study group by chance (like flipping a coin). You will be randomly put in one of the two study groups. You will have an equal chance of being placed in one of the groups shown below. A computer will randomly put you in a study group. We do this because no one knows if the results in one study group will be different than the other. The results could be better, the same or worse than the results in the other group. Once you are put in one group, you cannot switch to the other group. You and your doctor cannot choose the group you are in.

CSMC Date Effective: 1/28/2025

• **Single-blind:** This means that only the researchers will know which group you are in. They will not tell you which group you are in. Your physician will also not know which group you are in.

You can review the chart below to see what will happen during the study.



#### How long will you be in the study?

We think you will be in this study for about 8 weeks. This involves regular use of the VR program and weekly questionnaires.

About 1 month after completing the 8-week VR program, you may be invited to participate in a 1-hour Zoom interview. During this interview, a researcher will ask questions to better understand your experience with the VR program. You will receive a separate consent form for the interview closer to the end of the 8 weeks, if you are asked to take part in the interview.

#### 4. Possible Benefits From Taking Part in the Study

Being in this research study may or may not have direct medical benefit to you.

The possible benefits of taking part in the research study are reduction of abdominal pain and other IBS symptoms (e.g., bowel habit changes, bloating), and general improvement in mental health. Potential long-term benefits include continued improvement in abdominal pain and IBS symptoms, improved functionality, and improvements in overall physical and mental health. However, no benefit is guaranteed. It is possible that your condition may stay the same or even get worse.

We hope the information learned from this research study will contribute to societal knowledge about the safety and effectiveness of VR therapy among patients with IBS.

#### 5. Possible Risks and Discomforts of the Main Research Procedures

This section talks about the possible risks and discomforts of the main study procedures.

This study poses minimal risk to participants. Immediate risks may include minor psychological distress from questionnaire items asking about health and employment status.

CSMC Date Effective: 1/28/2025

There is also a small short-term risk of VR-related "cybersickness." Cybersickness is temporary feelings of vertigo, dizziness, nausea, headache, or feelings of anxiety. It usually resolves within minutes of removing the VR headset. Cybersickness has become less common with improvements in hardware and software. Technical advances have also reduced eye strain, minimized physical discomfort of wearing a VR headset, and reduced unnecessary visual motion, although the risk of these occurring is still present.

You may use glasses with the VR headset. With proper usage, the headset will not damage your glasses. Please follow usage instructions as the research team is not responsible for any damage to glasses that may occur from misuse of the equipment.

The Meta Quest 2 virtual reality headset weighs about 17.7 ounces (503 grams). Use of the headset can cause neck or back discomfort.

In rare instances, materials used in VR headsets have caused a mild rash which resolves when the VR headset is removed, and use is discontinued.

There are no anticipated long-term physical risks from participating in this study. There is a small risk of breach of confidentiality associated with the electronic collection and transmission of protected health information. This risk will be minimized by following proper procedures for assuring data integrity and confidentiality.

#### 6. Common Medical Procedures Performed for Research Purposes and Risks

The procedures listed below are often part of routine care for a person with your condition. They are not experimental procedures. That said, for this study these procedures and their risks are research-related. This means they are being *repeated* or performed *more frequently* for this study. These common procedures and their risks should be the same as when performed outside this study.

| Study Procedure | Related Risks |
|---|---|
| <b>Medications:</b> We will ask you about your | This does not have any physical risks. |
| past and current medications. Talk with the | |
| study team about any prescription drugs, | |
| over-the-counter drugs, supplements, and | |
| vitamins you take. | |
| <b>Demographic Information:</b> We will ask | This does not have any physical risks. |
| you about demographics, which may include | |
| your age, gender identity, race, and ethnicity. | |
| Screening of Depression: You will be | Tell the study team right away if you have feelings or |
| asked questions about your overall quality of | thoughts of harming yourself or others. This is so |
| life. This includes coping mechanisms or | that the study team can help you. The study team |
| times of depression. The study team may ask | will closely monitor your symptoms of depression. |
| you questions or ask you to answer | |
| questionnaires. | |

CSMC Date Effective: 1/28/2025

Questionnaires: You will be asked to complete questionnaires 10 times during the study (once after the consent call and once per week once you have received your VR headset). We will ask you questions to find out how you are feeling throughout the course of the study. We think it should take between 5-15 minutes to complete each questionnaire. Questionnaires will ask you to answer questions about your history with IBS, IBS symptoms, and bowel habits.

Some questions may make you feel uncomfortable or embarrassed.

The questionnaires will be labeled with a unique study number. This will allow only the research team can recognize you.

#### 7. Reasons Participation May Be Stopped by the Researcher or Sponsor

Your participation in this study may be stopped at any time. The researcher or the sponsor can stop your participation without your consent for any reason. If your participation is stopped early, the study doctor will discuss next steps with you. Some reasons for stopping your participation include:

- The study is stopped or suspended.
- Funding for the study is reduced, stopped, or withdrawn.
- It is in your best interest.
- You do not follow the study procedures.

#### 8. Voluntary Participation and Other Options

Taking part in research is voluntary. You have the right to choose not to take part. You can stop taking part in this research study at any time. You can do this without any penalty or loss of benefits to which you would be entitled outside of the study. Your choice not to take part or to stop taking part will not affect the care you get at Cedars-Sinai.

If you decide to stop taking part, we will keep any data collected on you up to the time you choose to stop. Also, if you stop taking part, the study team may ask you whether you want to give further data from your routine medical care.

You can decide not to take part in this study. You have other choices. For example, you may choose:

- To be treated following the usual clinical approach.
- To take part in a different study at Cedars-Sinai or elsewhere, if one is available.
- To not be treated.

The study team will discuss these options and their risks and benefits with you. You may also choose to discuss these with your treating physician.

CSMC Date Effective: 1/28/2025

#### 9. Confidentiality Protections

#### **General Confidentiality**

We will do our best to keep your personal information collected as part of this study private. But we cannot guarantee total privacy. We may put a copy of your research consent and authorization forms in your electronic medical record at Cedars-Sinai. Your personal information may be given out if required by law. Publications or presentations about this study at scientific meetings will not use your name and other identifiable personal information.

Organizations that may look at and/or copy your medical records for research oversight, quality assurance and data analysis include:

- Accrediting agencies (agencies that grant official certifications to educational institutions)
- Government and regulatory groups, such as the Food and Drug Administration (FDA) and Office for Human Research Protections (OHRP)
- The Institutional Review Board (IRB), which reviews research to protect people taking part in studies
- Safety monitors, which monitors the safety of individual participants and the overall safety of the study
- Companies that sponsor the study and authorized representatives of the sponsor

Attached to this consent form is an Authorization Form. It outlines with whom your information may be shared for this research and under what circumstances.

#### **Sharing Information**

We might share your information collected in this study. The information shared may include health data that could be used in future research. It might be shared with other researchers at Cedars-Sinai, other researchers outside of Cedars-Sinai, or third-party commercial entities for future research without additional informed consent from you. In some cases, your information may be submitted to a database or repository for future research. These databases and repositories have safeguards to prevent inappropriate access to and use of the information. Information that identifies you will be removed and will not be shared with other researchers or anyone outside of Cedars-Sinai. However, there is a remote possibility that someone could identify you.

#### **Clinical Trials Website**

A description of this clinical trial will be available on www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# **Protections From Forced Disclosures (Subpoenas) – Certificates of Confidentiality**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents or

CSMC Date Effective: 1/28/2025

samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence, unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate does not stop reporting that federal, state, or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases and threats to harm yourself or others. The Certificate cannot be used to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate does not stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also does not prevent your information from being used for other research, if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers, or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

#### 10. Research-Related Illness or Injury

#### **Contact in Case of Illness or Injury**

We do not expect you will have any illness or injury from this research study. If you believe that you are ill or have been injured from this study, please contact the study team at the phone number listed on page 1 of this consent form.

#### 11. Financial Considerations

#### **Costs of Participation**

You and your insurance company will not be charged for your participation in this research study.

#### **Payment**

You will be paid for participating in the research study. The total amount for completing the whole study is \$200. You will be paid within a week after meeting each milestone, see below.

The payment breakdown for this study is below:

- Milestone #1: After completing 3 out of the 4 weekly surveys (75%) in the 1st month of the study, you will be sent a \$100 Amazon gift code.
- Milestone #2: After completing 3 out of the 4 weekly surveys (75%) in the 2<sup>nd</sup> month of the study, and upon receipt of the VR headset by study staff, you will be sent a \$100 Amazon gift code.

CSMC Date Effective: 1/28/2025

Per Cedars-Sinai Medical Center policy, we will ask you to report the last 4 digits of your Social Security Number for tax purposes when distributing gift cards. The research team will not use this information for any other purposes other than payment.

You may have to fill out a W-9 form to get paid. Our accounting department at Cedars-Sinai will keep the W-9 form. Any amount of payment may be reportable to the IRS. If you receive \$600 or more from Cedars-Sinai in a calendar year, a 1099 form will be filed with the IRS in accordance with federal tax law. Check with a tax professional if you have questions.

If you are a Cedars-Sinai employee, you should provide your employee identification number to the research team. This allows your payment to be processed through Payroll. For your own protection and to comply with tax laws, your payment for taking part will be reported to the IRS together with other payment you get from Cedars-Sinai.

#### **Financial Interest in the Research**

A significant financial interest is a situation in which financial considerations could influence a person's professional judgment. This study has been designed to minimize the impact of the investigator's financial interest. You can ask the investigator to explain how the financial interest disclosed below will be managed.

The principal investigator, Christopher Almario, has no potential financial conflicts of interest with this study. Members of the research team, Brennan Spiegel (Co-Investigator) and Omer Liran (Co-Investigator), are co-founders of VRx Health, the company that developed and programmed the software being tested in this study.

Cedars-Sinai has a financial interest in this study. Under an Exclusive License Agreement with VRx Health, Cedars-Sinai holds a minority equity stake (approx. 2.5%) and will receive milestone, royalty, and annual maintenance fee payments.

#### 12. Contact for Questions or Problems

Please contact the investigator for questions, problems, or concerns about the research. Their contact information is on page 1 of this form.

You might have feedback, questions, problems, concerns or want to obtain more information about this study. If so, you can talk with someone who is not part of this study by contacting:

Cedars-Sinai Human Research Protection Program (HRPP)

Phone: 310-423-3783

Email: ResearchConcerns@cshs.org

Website: cedars-sinai.org/research/administration/office-of-research-compliance/review-

board.html

The Cedars-Sinai HRPP protects the rights and welfare of research participants.

CSMC Date Effective: 1/28/2025



## AUTHORIZATION FOR USE AND DISCLOSURE OF IDENTIFIABLE **HEALTH INFORMATION FOR RESEARCH** FOR CEDARS-SINAI AFFILIATED COVERED ENTITIES<sup>2</sup>

#### 1. USE AND DISCLOSURE OF HEALTH INFORMATION

If you agree to this Authorization, you give permission to the Sponsor, Principal Investigator, other investigators and their research team described in the Consent Form for Research ("Research Team") to use or disclose your identifiable health information ("private information") for the research study titled "Randomized controlled trial of virtual reality therapy for irritable bowel syndrome" which is described in the Consent Form for Research ("Consent Form") to which this Authorization is attached. In particular, you authorize the research team acting under the direction of the Principal Investigator to review your medical records and collect your private information from the following sources:

| ☐ Laboratory tests | ☐ Doctor/clinic records |
|---|---|
| ☐ Pathology reports | ☐ Hospital/medical records |
| ☐ Imaging reports (e.g., x-rays or scans) | ☐ Billing records |
| ☐ Photographs or videos of your image | |
| ■ Demographics, which may include, but is: | not limited to, age, gender identity, |
| race, ethnicity, and/or sexual orientation | |
| ☐ Mental health records | |
| ☐ Substance abuse records | |
| ☐ HIV test results | |
| ☑ Other tests or other types of medical inform | mation: survey responses |

#### 2. WHO WILL HAVE ACCESS TO YOUR PRIVATE INFORMATION?

Your private information will be used by and/or shared with the Research Team.

<sup>&</sup>lt;sup>2</sup> The Cedars-Sinai Affiliated Covered Entity ("ACE") is comprised of covered entities under the common ownership or control of Cedars-Sinai Health System, including Cedars-Sinai Medical Center (CSMC); Cedars-Sinai Medical Care Foundation; Cedars-Sinai Marina Del Rey Hospital (MDRH); Torrance Memorial Medical Center (TMMC); Torrance Health Association, Inc., d/b/a Torrance Memorial Physician Network; Huntington Hospital (HH), and Huntington Medical Foundation.

CSMC Date Effective: 1/28/2025

In addition to the research team, if applicable, the following parties may receive your private information and inspect your records:

- The reviewing Institutional Review Boards and Cedars-Sinai offices with authority to oversee research compliance.
- U.S. government agencies, such as the Food and Drug Administration and the Department of Health and Human Services.
- Researchers at other organizations who are participating in this research study.
- The Study Sponsor, its business partners, and Cedars-Sinai's business partners for matters related to research study oversight, conduct of the research, data analysis, use of research results in product development, and payment or reimbursement.
- Representatives from regulatory agencies in other countries may join in the review of your research records, including research-related medical reports and information, with the Sponsor and/or the FDA.

Cedars-Sinai takes steps to protect your private information when sharing it with the recipients described above. Though these steps and applicable law are meant to protect your private information, there is a risk that a recipient could share your private information without your permission.

# 3. WHEN WILL MY AUTHORIZATION EXPIRE?

By signing this document, you authorize the use and sharing of your private information until the end of the research study and any related optional sub-study you choose to participate in.

#### 4. REVOKING AUTHORIZATION

You may change your mind and revoke (take back) this Authorization at any time. Even if you revoke this Authorization, the research team may still use or disclose private information they already have obtained about you as necessary to maintain the integrity or reliability of the current research. To revoke this Authorization, you must write to the Principal Investigator of the research study by writing to the Office of Research Compliance and Quality Improvement, 6500 Wilshire Blvd, Suite 1800, Los Angeles, Calif. 90048 and/or emailing to ResearchConcerns@cshs.org.

#### 5. NOTICE OF RIGHTS AND OTHER INFORMATION

You do not have to agree to this Authorization, but if you do not agree, you may not participate in the research study. Cedars-Sinai may not condition (withhold or refuse) the provision of standard of care treatment for you on whether you agree to this Authorization.

If you agree to this Authorization, please sign on the appropriate signature line on the Signature Page. You will receive a copy of this Authorization.

CSMC Date Effective: 1/28/2025



# **Experimental Subject's Bill of Rights**

In accordance with California Health and Safety Code 24172, any person who is required to consent to participate as a subject in a research study involving a medical experiment or who is requested to consent on behalf of another has the right to:

- 1. Be informed of the nature and purpose of the experiment.
- 2. Be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized.
- 3. Be given a description of any attendant discomforts and risks to the subject reasonably to be expected from the experiment.
- 4. Be given an explanation of any benefits to the subject reasonably to be expected from the experiment, if applicable.
- 5. Be given a disclosure of any appropriate alternative procedures, drugs or devices that might be advantageous to the subject, and their relative risks and benefits.
- 6. Be informed of the avenues of medical treatment, if any, available to the subject after the experiment if complications should arise.
- 7. Be given an opportunity to ask any questions concerning the experiment or the procedure involved.
- 8. Be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation in the medical experiment without prejudice.
- 9. Be given a copy of any signed and dated written consent form used in relation to the experiment.
- 10. Be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion, or undue influence on the subject's decision.

CSMC Date Effective: 1/28/2025

# Signature Page

#### **Consent Form for Research and Authorization** for Use and Disclosure of Identifiable Health Information (Research)

If you agree to take part in this study, you should sign and date on the signature lines below. You will be given a signed and dated copy of this form. This includes the "Experimental Subject's Bill of Rights," "Authorization for Use and Disclosure of Identifiable Health Information (Research)" and any optional sub-study descriptions, when applicable.

#### Signature by the Participant

Main Research Study: I agree to take part in the research study described to me during the informed consent process and described in this informed consent form. My questions have been answered to my satisfaction.

| You will be given a signed and da | ted copy of this form | 1. |
|---|---|---|
| Participant name (please print) | Signature | Date |
| <b>Signature by the participant's pa</b> By providing my signature, I give perm below, in the research study described | nission for the participa | tion of my child, named |
| Name of Child (Print) | | |
| Parent/Guardian Name (Print) | Signature | Date of Signature |
| Authorization for Use and D<br>Information (Research): I he<br>information may be used and/or<br>"Authorization for Use and Disc<br>(Research)." | ereby agree that my<br>r disclosed in accord | identifiable health<br>lance with the |
| Participant name (please print) | Signature | Date |

CSMC IRB No: STUDY00003343 / MOD00011345 CSMC Date Effective: 1/28/2025

> (If applicable) Parent/Guardian Authorization for Use and Disclosure of Identifiable Health Information (Research): I hereby agree that my child's identifiable health information may be used and/or disclosed in accordance with this "Authorization for Use and Disclosure of Identifiable Health Information (Research)" form.

| Parent/Guardian Name (Print) | Signature | Date Signed |
|---|---|---|
| Signature by the Investigator I attest that all the elements of informed discussed fully in non-technical terms a questions asked by the participant were | vith the participant | t. I further attest that all |
| Investigator name (please print) | Signature | Date |
| Witness (Signature of a witness is required whe determined to have capacity to consent form, but choses to indicate via a "mark The witness signs the consent form to c that the individual verbally consented to | t is unable to read o<br>k" or verbally that l<br>onfirm that an oral | or physically sign the consent<br>he/she agrees to participate.<br>I consent process occurred, and |
| Witness name (please print) | Signature | Date |

CSMC Date Effective: 5/13/2025



# **CONSENT FORM FOR RESEARCH**For Cedars-Sinai and Participating Affiliates<sup>1</sup>

**Study title:** Randomized controlled trial of virtual reality therapy for irritable bowel syndrome.

**Sub-study title:** Interview for understanding IBS patient experience with SynerGI program

**Sponsor:** National Institute of Diabetes and Digestive and Kidney Diseases

Cedars-Sinai Principal Investigator: Christopher V. Almario, MD, MSHPM

Cedars-Sinai study contact phone number: 310-423-5434

- 1. Key Information
- 2. Purpose of the Sub-Study
- 3. Sub-Study Procedures
- 4. Possible Benefits From Taking Part in the Sub-Study
- 5. Possible Risks and Discomforts of the Main Research Procedures
- 6. Reasons Participation May Be Stopped by the Researchers or Sponsor
- 7. Voluntary Participation and Other Options
- 8. Confidentiality Protections
- 9. Research-Related Illness or Injury
- 10. Financial Considerations
- 11. Contact for Ouestions or Problems

Authorization for Use or Disclosure of Identifiable Health Information for Research

Signature Page

# 1. Key Information

Thank you for considering research participation. Research helps make medical and scientific advancements possible. In this form, we are asking for your consent to take part in this research study. Taking part in this research study is voluntary.

<sup>&</sup>lt;sup>1</sup> The **Cedars-Sinai Affiliated Covered Entity ("ACE")** is comprised of covered entities under the common ownership or control of Cedars-Sinai Health System, including Cedars-Sinai Medical Center (CSMC); Cedars-Sinai Medical Care Foundation; Cedars-Sinai Marina Del Rey Hospital (MDRH); Torrance Memorial Medical Center (TMMC); Torrance Health Association, Inc., d/b/a Torrance Memorial Physician Network; Huntington Hospital (HH), and Huntington Medical Foundation.

CSMC Date Effective: 5/13/2025

This section provides key information about the study. Please take your time to read this entire form. Also, please ask questions before deciding whether to take part in this research study. You are welcome to talk with family, friends and other healthcare providers before you decide.

- **Purpose:** The purpose of this sub-study is to get participant feedback on your IBS symptoms and the SynerGI program that you used for the main virtual reality (VR) study. Section 2 includes more details.
- **Procedures:** The main things that will happen in this sub-study are: you will be scheduled for a one-hour Microsoft Teams interview with a Cedars-Sinai study team member about a month after completing your participation in the virtual reality study. Section 3 includes more details.
- **Benefits:** You are not likely to be directly helped from being in this sub-study. But the information learned from this sub-study may help others in the future. Section 4 includes more details.
- **Risks:** All research studies involve some risks. Risks or discomforts from this sub-study may be: minor psychological distress from questions regarding IBS symptoms and health status. Section 5 includes more details.
  - o If you have problems during the sub-study, contact the study team using the contact information on the first page of this consent form.
- **Alternatives:** You can choose not to be in the sub-study.
- **New Information:** During the sub-study, we may find out new information about this sub-study. We will tell you about any important changes or new findings that may impact your decision to continue taking part in the sub-study.

### 2. Purpose of the Sub-Study

We are conducting interviews to hear from past participants from the randomized controlled trial of virtual reality therapy for irritable bowel syndrome study about their experiences with the SynerGI program and the impact it may have had on their IBS during the 8-week study. These interviews will be one-on-one with a study team member, and will take place virtually online using HIPAA-compliant, secure Microsoft Teams web conferencing software.

You are being asked to take part in this research study because you recently completed the randomized controlled trial of virtual reality therapy for irritable bowel syndrome study and were provided with the SynerGI program.

The sub-study will include up to 30 people in total.

CSMC Date Effective: 5/13/2025

#### 3. Sub-study Procedures

#### **Description of research procedures:**

- Interview: You will be asked to provide your experiences with IBS and your opinions on the SynerGI program.
  - o The interview will occur virtually, via Microsoft Teams. A Microsoft Teams link will be provided by the study team prior to the interview.
  - o The interview will be one-on-one with a study staff member, but there may be another staff member in the Microsoft Teams room to assist with notetaking.
  - You will be allowed to respond to questions or share other feedback you find relevant to your experiences in the study, with the VR headset and program and any impact on your IBS. If you feel uncomfortable or embarrassed answering any question, you may choose to not answer it.
  - o The interview should take about 60 minutes to complete.
  - Video recordings will be made during the interview and will only be used for transcription purposes, meaning that we will listen to the audio, write down everything that was said, and assign quotes to a unique ID that will mask your identity.
  - The recordings will be destroyed after being transcribed. Neither the recordings nor the transcription will be reproduced or published in any other format or setting.

#### How long will you be in the sub-study?

We think you will be in this sub-study for about 60 minutes.

### 4. Possible Benefits From Taking Part in the Sub-Study

You should not expect to benefit from taking part in this sub-study. We don't expect any direct benefit to you from being in the sub-study.

We hope the information learned from this sub-study will help identify areas of improvement for the SynerGI program and how it relates to your IBS. This information can help researchers improve the programming so that it can better help patients with IBS in the future.

#### 5. Possible Risks and Discomforts of the Research Procedures

This section talks about the possible risks and discomforts of the study procedures.

• **Interview:** There are no physical risks to you expected from taking part in this substudy. It is possible that some of the items discussed during the interview may make you feel uncomfortable or embarrassed. You are not required to respond to any item that you do not wish to answer. If any question makes you feel uncomfortable, you can simply tell the interviewer you wish to pass on answering the question. This will not affect your participation in the study. There is also a risk of loss of confidentiality of records; however, there are procedures in place to minimize this risk. For example, any

CSMC Date Effective: 5/13/2025

transcripts or notes taken during the interview will not include your name or identifying information.

#### 6. Reasons Participation May Be Stopped by the Researcher or Sponsor

Your participation in this sub-study may be stopped at any time. The researcher or the sponsor can stop your participation without your consent for any reason. If your participation is stopped early, the researcher will discuss next steps with you. Some reasons for stopping your participation include:

- The sub-study is stopped or suspended.
- Funding for the sub-study is reduced, stopped or withdrawn.
- It is in your best interest.
- You do not follow the sub-study procedures.

#### 7. Voluntary Participation and Other Options

Taking part in research is voluntary. You have the right to choose not to take part. You can stop taking part in this research sub-study at any time. You can do this without any penalty or loss of benefits to which you would be entitled outside of the sub-study. Your choice not to take part or to stop taking part will not affect the care you get at Cedars-Sinai.

If you decide to stop taking part, we will keep any data collected on you up to the time you choose to stop. Also, if you stop taking part, the study team may ask you whether you want to give further data from your routine medical care.

### 8. Confidentiality Protections

#### **General Confidentiality**

We will do our best to keep your personal information collected as part of this sub-study private. But we cannot guarantee total privacy. We may put a copy of your research consent and authorization forms in your electronic medical record at Cedars-Sinai. Your personal information may be given out if required by law. Publications or presentations about this study at scientific meetings will not use your name and other identifiable personal information.

Organizations that may look at and/or copy your medical records for research oversight, quality assurance and data analysis include:

- Accrediting agencies (agencies that grant official certifications to educational institutions)
- Government and regulatory groups, such as the Food and Drug Administration (FDA) and Office for Human Research Protections (OHRP)
- The Institutional Review Board (IRB), which reviews research to protect people taking part in studies
- Safety monitors, which monitor the safety of individual participants and the overall safety of the study
- Companies that sponsor the study and authorized representatives of the sponsor

CSMC Date Effective: 5/13/2025

Attached to this consent form is an Authorization Form. It outlines with whom your information may be shared for this research and under what circumstances.

#### **Sharing Information**

We might share your information collected in this study. The information shared may include health data that could be used in future research. It might be shared with other researchers at Cedars-Sinai, other researchers outside of Cedars-Sinai, or third-party commercial entities for future research without additional informed consent from you. In some cases, your information may be submitted to a database or repository for future research. These databases and repositories have safeguards to prevent inappropriate access to and use of the information. Information that identifies you will be removed and will not be shared with other researchers or anyone outside of Cedars-Sinai. However, there is a remote possibility that someone could identify you.

#### **Clinical Trials Website**

A description of this clinical trial will be available on www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# Protections From Forced Disclosures (Subpoenas) – Certificates of Confidentiality

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence, unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate does not stop reporting that federal, state, or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases and threats to harm yourself or others. The Certificate cannot be used to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate does not stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also does not prevent your information from being used for other research, if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers, or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

CSMC Date Effective: 5/13/2025

### 9. Research-Related Illness or Injury

#### **Contact in Case of Illness or Injury**

We do not expect you will have any illness or injury from this research sub-study. If you believe that you are ill or have been injured from this sub-study, please contact the study team at the phone number listed on page 1 of this consent form.

#### 10. Financial Considerations

#### **Costs of Participation**

You and your insurance company will not be charged for your participation in this sub-study.

#### **Payment**

You will be paid for completing the interview with a study team member. The total amount for completing the interview is \$100. You will be paid after the interview has been completed.

You may have to fill out a W-9 form to get paid. Our accounting department at Cedars-Sinai will keep the W-9 form. Any amount of payment may be reportable to the IRS. If you receive \$600 or more from Cedars-Sinai in a calendar year, a 1099 form will be filed with the IRS in accordance with federal tax law. Check with a tax professional if you have questions.

If you are a Cedars-Sinai employee, you should provide your employee identification number to the research team. This allows your payment to be processed through Payroll. For your own protection and to comply with tax laws, your payment for taking part will be reported to the IRS together with other payment you get from Cedars-Sinai.

#### **Financial Interest in the Research**

A significant financial interest is a situation in which financial considerations could influence a person's professional judgment. This sub-study has been designed to minimize the impact of the investigator's financial interest. You can ask the investigator to explain how the financial interest disclosed below will be managed.

The principal investigator, Christopher Almario, has no potential financial conflicts of interest with this study. Members of the research team, Brennan Spiegel (Co-Investigator) and Omer Liran (Co-Investigator), are co-founders of VRx Health, the company that developed and programmed the software being tested in this study.

Cedars-Sinai has a financial interest in this study. Under an Exclusive License Agreement with VRx Health, Cedars-Sinai holds a minority equity stake (approx. 2.5%) and will receive milestone, royalty, and annual maintenance fee payments.

#### 11. Contact for Questions or Problems

Please contact the investigator for questions, problems or concerns about the research. Their contact information is on page 1 of this form.

CSMC Date Effective: 5/13/2025

You might have feedback, questions, problems, concerns or want to obtain more information about this study. If so, you can talk with someone who is not part of this study by contacting:

Cedars-Sinai Human Research Protection Program (HRPP)

Phone: 310-423-3783

Email: ResearchConcerns@cshs.org

Website: cedars-sinai.org/research/administration/office-of-research-compliance/review-

board.html

The Cedars-Sinai HRPP protects the rights and welfare of research participants.

CSMC Date Effective: 5/13/2025



### AUTHORIZATION FOR USE AND DISCLOSURE OF IDENTIFIABLE HEALTH INFORMATION FOR RESEARCH FOR CEDARS-SINAI AFFILIATED COVERED ENTITIES<sup>2</sup>

#### 1. USE AND DISCLOSURE OF HEALTH INFORMATION

If you agree to this Authorization, you give permission to the Sponsor, Principal Investigator, other investigators and their research team described in the Consent Form for Research ("Research Team") to use or disclose your identifiable health information ("private information") for the research study titled "Interview for understanding IBS patient experience with SynerGI program" which is described in the Consent Form for Research ("Consent Form") to which this Authorization is attached. In particular, you authorize the research team acting under the direction of the Principal Investigator to review your medical records and collect your private information from the following sources:

| ☐ Laboratory tests ☐ Pathology reports ☐ Imaging reports (e.g., x-rays or scans) | <ul><li>☐ Doctor/clinic records</li><li>☐ Hospital/medical records</li><li>☐ Billing records</li></ul> |
|---|---|
| ☐ Photographs or videos of your image | |
| ■ Demographics, which may include, but it | is not limited to, age, gender identity, |
| race, ethnicity, and/or sexual orientation | |
| ☐ Mental health records | |
| <ul><li>☐ Substance abuse records</li><li>☐ HIV test results</li></ul> | |
| ☑ Other tests or other types of medical info | ormation: interview responses |

#### 2. WHO WILL HAVE ACCESS TO YOUR PRIVATE INFORMATION?

Your private information will be used by and/or shared with the Research Team.

<sup>&</sup>lt;sup>2</sup> The Cedars-Sinai Affiliated Covered Entity ("ACE") is comprised of covered entities under the common ownership or control of Cedars-Sinai Health System, including Cedars-Sinai Medical Center (CSMC); Cedars-Sinai Medical Care Foundation; Cedars-Sinai Marina Del Rey Hospital (MDRH); Torrance Memorial Medical Center (TMMC); Torrance Health Association, Inc., d/b/a Torrance Memorial Physician Network; Huntington Hospital (HH), and Huntington Medical Foundation.

CSMC Date Effective: 5/13/2025

In addition to the research team, if applicable, the following parties may receive your private information and inspect your records:

- The reviewing Institutional Review Boards and Cedars-Sinai offices with authority to oversee research compliance.
- U.S. government agencies, such as the Food and Drug Administration and the Department of Health and Human Services.
- Researchers at other organizations who are participating in this research study.
- The Study Sponsor, its business partners, and Cedars-Sinai's business partners for matters related to research study oversight, conduct of the research, data analysis, use of research results in product development, and payment or reimbursement.
- Representatives from regulatory agencies in other countries may join in the review of your research records, including research-related medical reports and information, with the Sponsor and/or the FDA.

Cedars-Sinai takes steps to protect your private information when sharing it with the recipients described above. Though these steps and applicable law are meant to protect your private information, there is a risk that a recipient could share your private information without your permission.

#### 3. WHEN WILL MY AUTHORIZATION EXPIRE?

By signing this document, you authorize the use and sharing of your private information until the end of the research study and any related optional sub-study you choose to participate in.

#### 4. REVOKING AUTHORIZATION

You may change your mind and revoke (take back) this Authorization at any time. Even if you revoke this Authorization, the research team may still use or disclose private information they already have obtained about you as necessary to maintain the integrity or reliability of the current research. To revoke this Authorization, you must write to the Principal Investigator of the research study by writing to the Office of Research Compliance and Quality Improvement, 6500 Wilshire Blvd, Suite 1800, Los Angeles, Calif. 90048 and/or emailing to ResearchConcerns@cshs.org.

#### 5. NOTICE OF RIGHTS AND OTHER INFORMATION

You do not have to agree to this Authorization, but if you do not agree, you may not participate in the research study. Cedars-Sinai may not condition (withhold or refuse) the provision of standard of care treatment for you on whether you agree to this Authorization.

CSMC Date Effective: 5/13/2025

If you agree to this Authorization, please sign on the appropriate signature line on the Signature Page. You will receive a copy of this Authorization.

# Signature Page

#### **Consent Form for Research and Authorization** for Use and Disclosure of Identifiable Health Information (Research)

If you agree to take part in this study, you should sign and date on the signature lines below. You will be given a signed and dated copy of this form. This includes the "Experimental Subject's Bill of Rights," "Authorization for Use and Disclosure of Identifiable Health Information (Research)" and any optional sub-study descriptions, when applicable.

#### Signature by the Participant

**Main Research Study:** I agree to take part in the research study described to me during the informed consent process and described in this informed consent form. My questions have been answered to my satisfaction.

| Participant name (please print) | Signature | Date |
|---|---|---|
| <b>Authorization for Use and Di Information (Research):</b> <i>I he information may be used and/or</i> | reby agree that my | identifiable health |
| "Authorization for Use and Discl<br>(Research)." | | |

I attest that all the elements of informed consent described in this form have been discussed fully in non-technical terms with the participant. I further attest that all questions asked by the participant were answered to the best of my knowledge.

Signature Investigator name (please print) Date **Interpreter/Witness** (Signature of an interpreter is only required when enrolling a non-English-speaking subject with the assistance of an interpreter and IRB-approved "short form" consent processes. The witness may be any person who is conversant in both English and the language of the non-English-speaking subject, such as a certified hospital interpreter, study staff, a family member or other person. The witness signs the consent forms to confirm that the oral interpretation occurred. Signature of a witness is required when an English-speaking subject who has been determined to have capacity to consent is unable to read or physically sign the consent form but chooses to indicate via a "mark" or verbally that he/she agrees to participate. The witness signs the consent form to confirm that an oral consent process occurred and that the individual verbally consented to participate in the research.)

CSMC IRB No: STUDY00003343 / MOD00012031

Interpreter/Witness name (please print) Signature

CSMC Date Effective: 5/13/2025

Date of signature